CLINICAL TRIAL: NCT02584725
Title: Determining the Optimal Dose of Tranexamic Acid in Decreasing Blood Loss During Lower Extremity Total Joint Arthroplasty
Brief Title: Tranexamic Acid Dosing for Total Joint Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Robert Maniker, Assistant Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAM9601
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee
Keywords: Tranexamic Acid; Total Joint Arthroplasty; Intraoperative Blood Loss
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg/kg/dose tranexamic acid (Active Comparator): 5 mg/kg tranexamic acid IV, administered twice, once 20 minutes prior to surgical incision and once at when surgical wound closure begins
  Interventions: Drug: Tranexamic Acid
- 10 mg/kg/dose tranexamic acid (Active Comparator): 10 mg/kg tranexamic acid IV, administered twice, once 20 minutes prior to surgical incision and once at when surgical wound closure begins
  Interventions: Drug: Tranexamic Acid
- 15 mg/kg/dose tranexamic acid (Active Comparator): 15 mg/kg tranexamic acid IV, administered twice, once 20 minutes prior to surgical incision and once at when surgical wound closure begins
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Comparison of 3 different doses of the drug
  Other Names: Lysteda

SUMMARY:
The purpose of this study is to determine the effect of increasing doses of tranexamic acid (TXA) on limiting blood loss during total knee and total hip arthroplasty as defined by a change in hemoglobin from pre-operative baseline to the first post-operative day.

DETAILED DESCRIPTION:
The study is a prospective, randomized, double-blinded trial comparing three different doses of TXA (5mg/kg, 10mg/kg, 15mg/kg) in decreasing blood loss during and after total knee and total hip arthroplasty. Patients undergoing total knee arthroplasty and total hip arthroplasty will be analyzed separately, in sub-group analysis. The primary endpoint will be the change in hemoglobin from baseline to the first post-operative day (POD#1).

Patients will initially be identified by their orthopedic surgeon if they meet the inclusion and exclusion criteria. They will be informed about the study and provided with the consent form in the office, which they will be able to review further prior to the date of surgery. If the patient wishes to participate, formal written consent will be completed by one of the study investigators or a member of the regional anesthesia team. Patients will then be randomized to one of three groups. The anesthesia team responsible for the subject patient's care will receive two twenty milliliter syringes of medication. The syringe labeled "Study medication #1" will be administered intravenously over 20 minutes beginning at the start of surgical skin preparation, and the syringe labeled "Study medication #2" will be administered over 20 minutes beginning at the start of surgical wound closure. The syringes for group 1 (low-dose TXA) will each contain 5mg/kg TXA, diluted to 20 milliliters with saline. The syringes for group 2 (moderate-dose TXA) will each contain 10mg/kg TXA, diluted to 20 milliliters with saline. The syringes for group 3 (high-dose TXA) will each contain 15mg/kg TXA, diluted to 20 milliliters with saline. The anesthesia team will document the total intra-operative estimated blood loss as well as the amount of blood in the suction canister at the end of the surgery (as calculated by volume in the suction bucket minus volume of irrigation used).

The intraoperative course will be standardized for all patients included in the study. For total knee arthroplasty patients, the anesthesia will consist of a long-acting femoral or adductor canal peripheral nerve block, followed by a standardized spinal anesthetic using 15mg of plain isobaric bupivacaine. For total hip arthroplasty patients, the anesthesia will consist of a standardized spinal anesthetic using 15mg of plain isobaric bupivacaine. In those patients for whom spinal anesthesia is contraindicated or refused, general anesthesia will be performed and these patients will be excluded from the study. All patients initially enrolled, but excluded secondary to administration of a general anesthetic will be analyzed via an intention-to-treat method. Administration of intravenous crystalloid solutions will be per the discretion of the anesthesia team participating in the intra-operative portion of each patient's care, and will be documented for purposes of this study by the anesthesia team.

On PODs #0, #1 and #2, all patients will undergo standard post-operative blood work which includes a complete blood count. When working with physical therapy on POD#1 and POD#2, assessment of ability to sit, stand, and walk (yes/no) will be recorded. Assessment of pain scores via a VAS (0-10 scale, with 0 being no pain and 10 being the worst 05/26/2016 pain) will be recorded on POD#1 and POD#2. Assessment of subjective sense of overall wellbeing (a 0-10 scale, with 0 being the worst patients have ever felt, and 10 representing pre-operative baseline) will be recorded on POD #1 and #2. Patients will also be monitored via clinical exam for incidence of seizure, transient ischemic attack, stroke, myocardial infarction, deep venous thrombosis, and pulmonary embolus in the first 48 post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total knee arthroplasty or primary unilateral total hip arthroplasty under spinal anesthesia at Columbia University Medical Center/ New York Presbyterian Hospital.

Exclusion Criteria:

* Non-English speaking.
* Patient refusal to participate.
* Weight exceeding 100kg.
* Baseline hemoglobin of less than 10.
* Repeat, revision, or bilateral surgery.
* Known sensitivity or allergy to Tranexamic Acid.
* Active intra-vascular clotting.
* History of coagulopathy or congenital thrombophilia.
* Thromboembolic event in the 12 months prior to enrollment.
* Percutaneous coronary intervention requiring a drug eluting stent in the 12 months prior to enrollment.
* History of anticoagulant medication use unless stopped prior to surgery as recommended by and in accordance with the American Society of Regional Anesthesia Guidelines.
* Use of a general anesthetic in the current anesthetic.
* Blood transfusion for a hemoglobin value which deviates from the study's transfusion protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maniker, MD, Principal Investigator — Columbia University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Started | 28 | 28 | 28
Completed | 28 | 28 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid | Total
Number analyzed (Participants) | 28 | 28 | 28 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 12 | 30
  >=65 years | 18 | 20 | 16 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 20 | 59
  Male | 6 | 11 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin From Baseline to the First Post-operative Day (POD#1)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
g/dl | 2.15 (1.19) | 2.06 (0.81) | 2.11 (0.97)

2. Secondary Outcome: Change in Hemoglobin From Baseline to POD#0
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
g/dL | 1.34 (1.19) | 1.30 (0.71) | 1.16 (0.94)

3. Secondary Outcome: Change in Hemoglobin From Baseline to POD#2
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
g/dL | 2.50 (1.2) | 2.59 (0.67) | 2.28 (1.1)

4. Secondary Outcome: Number of Participants Requiring Blood Transfusion From the Intra-operative Period Into the End of POD#2
Description: Number or count of participants requiring transfusion.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
Participants | 1 | 0 | 0

5. Secondary Outcome: Total Estimated Intra-operative Blood Loss
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
mL | 321.43 (276.21) | 322.32 (261.84) | 376.25 (314.08)

6. Secondary Outcome: Volume of Blood in the Surgical Suction Canister at the End of Surgery
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
mL | 282.50 (262.19) | 283.93 (240.31) | 329.11 (285.89)

7. Secondary Outcome: Count of Participants Able to Sit on Post-Operative Day 1 (POD1) and Post-Operative Day 2 (POD2)
Description: Count of participants able to sit on POD1 and POD2 as assessed by a mobility assessment.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
Participants
  Count of Participants Able to Sit POD1 | 26 | 28 | 28
  Count of Participants Able to Sit POD2 | 27 | 28 | 28

8. Secondary Outcome: Count of Participants Able to Stand on POD1 and POD2
Description: Count of participants able to stand on POD1 and POD2 as assessed by a mobility assessment.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
Participants
  Count of Participants Able to Stand POD1 | 25 | 28 | 27
  Count of Participants Able to Stand POD2 | 28 | 28 | 28

9. Secondary Outcome: Count of Participants Able to Walk on POD1 and POD2
Description: Count of participants able to Walk on POD1 and POD2 as assessed by a mobility assessment.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
Participants
  Count of Participants Able to Walk POD1 | 26 | 28 | 25
  Count of Participants Able to Walk POD2 | 28 | 28 | 28

10. Secondary Outcome: Visual Analog Scale (VAS) Pain Scores on POD#1 and POD#2
Description: The VAS measures pain on a scale of 0-10, with 0=no pain and 10=worst possible pain.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
score on a scale
  VAS Pain Score POD#1 | 5.18 (2.76) | 3.82 (2.98) | 4.36 (2.23)
  VAS Pain Score POD#2 | 4.63 (2.62) | 3.89 (2.69) | 4.32 (2.09)

11. Secondary Outcome: Wellbeing Questionnaire Score on POD#1 and POD#2
Description: Patients' self-reported scores on a scale of overall feeling of wellbeing on POD#1 and POD#2. Scores range from 0-10, with 0= "worst I have ever felt" and 10= "feel just as well as before surgery."
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
score on a scale
  Wellbeing Score POD#1 | 6.54 (2.91) | 7.71 (2.62) | 7.04 (2.25)
  Wellbeing Score POD#2 | 7.15 (2.96) | 8.04 (2.08) | 7.39 (2.13)

12. Secondary Outcome: Count of Seizure, Transient Ischemic Attack, Stroke, Myocardial Infarction, Deep Venous Thrombosis, and Pulmonary Embolus
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
Number analyzed (Participants) | 28 | 28 | 28
participants
  Post-operative Seizure | 0 | 0 | 0
  Post-operative Transient Ischemic Attack | 0 | 0 | 0
  Post-operative Myocardial Infarction | 0 | 0 | 0
  Post-operative Deep Vein Thrombosis | 0 | 0 | 0
  Post-operative Pulmonary Embolus | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 2 Days
Description: Monitoring of potential adverse events will be done via clinical exam in the first 48 hours post-operatively. The definition of adverse event does not differ from the ClinicalTrials.gov definition.
Arm/Group | 5 mg/kg/Dose Tranexamic Acid | 10 mg/kg/Dose Tranexamic Acid | 15 mg/kg/Dose Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg/Dose Tranexamic Acid (N=28) | 10 mg/kg/Dose Tranexamic Acid (N=28) | 15 mg/kg/Dose Tranexamic Acid (N=28)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT02584725/Prot_SAP_000.pdf